CLINICAL TRIAL: NCT00265005
Title: Dose-Ranging, Safety And Efficacy Of Cathflo(TM) Activase(R) (Alteplase) For The Treatment Of Central Catheter Occlusion In Neonates And Infants; Phase I
Brief Title: Safety and Efficacy of Tissue Plasminogen Activator (tPA) in Neonates and Infants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: difficulty in recruiting subjects
Sponsor: University of Louisville (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Janice E. Sullivan, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tPA 255-04
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2015-12

CONDITIONS: Thrombosis
Keywords: alteplase; occluded central venous catheter; occluded arterial catheter; occluded PICC; neonates; infants
MeSH Terms: conditions — Thrombosis | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All (Experimental): All subjects receive active drug up to a total of 3 doses
  Interventions: Drug: alteplase

INTERVENTIONS:
Drug: alteplase — Iv administration of 1 mg/ml up to two times and 2 mg/ml if needed.
  Other Names: Cathflo Activase

SUMMARY:
The purpose of this study is to determine if alteplase is effective in dissolving a clot in a catheter in a large vein (central venous line or PICC line) or artery in infants less than 6 months of age.

DETAILED DESCRIPTION:
Hospitalized patients with central access devices will be screened. Ninety subjects with at least one occluded lumen of a central access device will be eligible. Thirty subjects will be enrolled in each of the following age groups: 28-<34 weeks CGA, 34- < 40 weeks CGA, and 40 weeks to 66 weeks CGA.

Inclusion Criteria

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent by the parent or legal guardian and comply with study assessments for the full duration of the study.
* Hospitalized premature neonates (28-< 34 weeks CGA), term neonates (34-<40 weeks CGA) and infants (40 weeks to 66 weeks CGA).
* Presence of a central access device. All types of permanent and temporary catheters are eligible [e.g., central venous catheter (CVC), peripherally-inserted central catheter (PICC), umbilical arterial catheter (UAC), or umbilical venous catheter (UVC)] except hemodialysis catheters. The catheter must be properly inserted as evidenced by the ability to have used the catheter at least once for its intended purpose (i.e., to withdraw blood and/or infuse fluids) and documentation of correct catheter placement radiographically within 48 hours of the catheter becoming non-patent.
* partial or total occlusion of at least one lumen of the catheter.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

* CGA > 66 weeks
* Incorrect catheter placement (see section 3.1) or evidence of mechanical occlusion
* By clinical examination there is evidence that the catheter has migrated or become dislodged. This is determined by confirming the depth to which the catheter had been positioned on insertion or adjusted to after placement.
* There is evidence of mechanical obstruction of the catheter on the portion (is any) that is visible from the catheter hub to the skin insertion site (e.g., kinking or twisting of the catheter).
* Occlusion due to suspected drug precipitate in the opinion of the investigator
* Active internal bleeding, involving intracranial and retroperitoneal sites, or the gastrointestinal, genitourinary, or respiratory tracts
* Recent history (i.e., < 6 months) of intraventricular hemorrhage (IVH) or other active intracranial process that could predispose to intracranial bleeding
* Superficial or surface bleeding, observed mainly at vascular puncture and access sites (e.g., venous cutdowns, arterial punctures) or site of recent surgical intervention
* Any of the following known or suspected hemorrhagic events within the preceding 7 days or any other significant bleeding risk:
* Gastrointestinal bleeding
* Intra-ocular surgery
* Any of the following known events or suspected hemorrhagic events within the preceding 48 hours
* Major surgery (excluding central line placement)
* Organ biopsy
* Major trauma
* Puncture of a non-compressible vessel within the previous 48 hours
* Treatment with indomethacin within the previous 48 hours
* Received any fibrinolytic agent within 24 hours of enrollment
* Known risk for embolization, including history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis, and subacute bacterial endocarditis
* Known hypersensitivity to Alteplase or any component in the formulation of CathfloTM Activase®
* Prior enrollment in the current study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated or the patient has a known condition for which bleeding constitutes a significant hazard
* Participation in another interventional investigation or trial within the previous 30 days
* Documented or suspected catheter infection
* Thrombocytopenia (i.e. platelet count < 20,000)

METHOD OF TREATMENT ASSIGNMENT This is an open-label study and all subjects will receive CathfloTM Activase.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent by the parent or legal guardian and comply with study assessments for the full duration of the study
* Hospitalized premature neonates (28- < 34 weeks CGA), term neonates (34 weeks-< 40 weeks CGA) and infants (> = 40 weeks to 6 months CGA).
* Presence of central access device. All types of permanent and temporary catheters are eligible [e.g., central venous catheter (CVC), peripherally-inserted central catheter (PICC), umbilical arterial catheter (UAC), or umbilical venous catheter (UVC)] except hemodialysis catheters. The catheter must be properly inserted as evidenced by the ability to have used the catheter at least once for its intended purpose (i.e., to withdraw blood and/or infuse fluids)and documentation correct catheter placement radiographically within 48 hours of the catheter becoming non-patent.
* Partial or total occlusion of at least one lumen of the catheter

Exclusion Criteria:

* CGA > 66 weeks
* Incorrect catheter placement or evidence of mechanical occlusion
* Occlusion due to suspected drug precipitate
* Active internal bleeding, involving intracranial or retroperitoneal sites, or the gastrointestinal, genitourinary, or respiratory tracts
* Recent history (i.e., < 6 months) of intraventricular hemorrhage (IVH) or other active intracranial process that could predispose to intracranial bleeding
* Superficial or surface bleeding, observed mainly at vascular puncture and access sites (e.g., venous cutdowns, arterial punctures) or site of recent surgical intervention
* Any of the following known or suspected hemorrhagic events within the preceding 7 days or any other significant bleeding risk:

  * Gastrointestinal bleeding
  * Intra-ocular surgery
* Any of the following known events or suspected hemorrhagic events within the preceding 48 hours

  * Major surgery (excluding central line placement)
  * Organ biopsy
  * Major trauma
* Puncture of a non-compressible vessel within the previous 48 hours
* Treatment with indomethacin within the previous 48 hours
* Received any fibrinolytic agent within 24 hours of enrollment
* Known risk for embolization, including history of left heart thrombus, mitral mitral stenosis with atrial fibrillation, acute pericarditis, and subacute bacterial endocarditis
* Known hypersensitivity to alteplase or any component in the formulation of CathfloTM Activase®
* Prior enrollment in the current study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated or the patient has a known condition for which bleeding constitutes a significant hazard
* Participation in another simultaneous interventional medical investigation or trial
* Documented or suspected catheter infection
* Thrombocytopenia (i.e. platelet count < 20,000)

Ages: 28 Weeks to 66 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Restoration of central access device patency following one, two or three instillations of t-PA. | within 180 minutes of administering the study drug

SECONDARY OUTCOMES:
Restoration of patency following instillation of 1 mg/mL (i.e., first instillation) | within 60 minutes from the first instillation of study drug
Restoration of patency following instillation of 1 mg/mL (i.e., second instillation) | within 60 minutes from the second instillation of study drug
Restoration of patency following instillation of 2 mg/mL (i.e., third instillation) | within 60 minutes from the third instillation of study drug
The following safety outcome measure will be evaluated: • Major bleeding complications • Sepsis • Embolic events • All serious adverse events | Within 14 days of study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Janice E Sullivan, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States